CLINICAL TRIAL: NCT04776928
Title: Testing a Provider-Level Feedback Intervention to Optimize Postoperative Prescribing - Aim 3 Phase 1
Brief Title: Testing a Provider-Level Feedback Intervention to Optimize Postoperative Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jennifer Waljee, Associate Professor of Surgery and Associate Professor of Orthopaedic Surgery, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUM00186352; 5R01DA042859-04 (NIH)
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Opioid Prescribing
Keywords: Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provider-level push report notifications (Experimental): Push reports will be sent via using a secure email client. The email will be sent to the email address provided to the study team by the surgeon or site.
  Interventions: Behavioral: Push reports
- No intervention (No Intervention): Sites who did not sign Exhibit B-1.

INTERVENTIONS:
Behavioral: Push reports — Surgeons in the experimental arm will receive provider-level push report notifications through an email displaying their personal prescribing performance compared to Michigan Opioid Prescribing Engagement Network (OPEN) prescribing guidelines and their de-identified peers.
  The push report will also include a link to the secure MSQC data platform that displays more information about the case so the surgeon can further investigate prescribing information. The email will also contain contact information for the study team so as to help any surgeons troubleshoot, learn more, request to stop receiving reports, etc.
  Arms: Provider-level push report notifications

SUMMARY:
The objective of this project is to leverage the Michigan Surgical Quality Collaborative's (MSQC) existing network and surgeon performance feedback platform to improve opioid prescribing practices for surgeons within the network found to be prescribing in a manner discordant with published guidelines and to inform best practices for future surgical quality improvement initiatives.

The study is being completed to learn more about the effectiveness, feasibility, and acceptability and that the goal is both to evaluate how effective this intervention and mechanism are for changing surgeon opioid prescribing behavior and to inform best practices for future quality initiatives. The study hypothesizes that provider-level feedback will allow clinicians to tailor postoperative prescribing more closely to patient consumption, and reduce excess postoperative prescribing.

The cohort of surgeons which have been identified as outliers by the Michigan Surgical Quality Collaborative (MSQC) will be be invited to participate in this trial. The study team will send surgeons belonging to sites that signed the Exhibit B-1 form the provider-level push notifications (98 participants). In this study de-identified prescribing data will also be analyzed for sites that do not sign the Exhibit B-1 form (105 participants).

The study team will approach 98 surgeons receiving the provider-level push notifications in one wave.

ELIGIBILITY:
Inclusion Criteria:

* Surgeons already participating in and sharing data with the Michigan Surgical Quality Collaborative (MSQC) who perform procedures of interest
* Surgeons within MSQC who have median prescribing > 1 pill equivalents over the published recommendation
* Surgeons within MSQC who perform surgeries at a hospital that have agreed to participate in this research

Exclusion Criteria:

* Surgeons not identified in the MSQC data as having a valid National Provider Identifier (NPI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer F Waljee, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Provider-level Push Report Notifications: Push reports will be sent via using a secure email client. The email will be sent to the email address provided to the study team by the surgeon or site.
  Push reports: Surgeons in the experimental arm will receive provider-level push report notifications through an email displaying their personal prescribing performance compared to Michigan Opioid Prescribing Engagement Network (OPEN) prescribing guidelines and their de-identified peers.
  The push report will also include a link to the secure MSQC data platform that displays more information about the case so the surgeon can further investigate prescribing information. The email will also contain contact information for the study team so as to help any surgeons troubleshoot, learn more, request to stop receiving reports, etc.
Period: Overall Study
Arm/Group | Provider-level Push Report Notifications | No Intervention
Started | 95 | 122
Completed | 95 | 122
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Provider-level Push Report Notifications | No Intervention | Total
Number analyzed (Participants) | 95 | 122 | 217
Age, Continuous [Mean (Standard Deviation); unit: Years] — Data on Age was not collected for participants. MSQC does not collect this data for surgeons. Population: Data on Age was not collected for participants (surgeon participant). MSQC does not collect this data for surgeons.
Sex: Female, Male [Count of Participants; unit: Participants] — Data on Sex was not collected for participants (surgeon participants). MSQC does not collect this data for surgeons. Population: Data on Sex was not collected for participants (surgeon participants). MSQC does not collect this data for surgeons.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 95 | 122 | 217
Prescribing Practices [Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)] — Results represent average number of opioid doses (measured in oral morphine equivalents or OMEs) prescribed by surgeon participants that exceed current guidelines of more than 1 pill (7.5 opioid oral morphine milligram equivalent or MMEs).
  Morphine Milligram Equivalents (MME) | 68.5 (56.87) | 64.3 (53.42) | 66.4 (55.21)

OUTCOME MEASURES:

1. Primary Outcome: Change in Opioid Prescribed Following the Intervention
Description: Oral morphine equivalents prescribed adjusted for surgery type as reported through MSQC data.
Time Frame: up to 5 months from enrollment
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Provider-level Push Report Notifications | No Intervention
Number analyzed (Participants) | 95 | 122
Morphine Milligram Equivalents (MME) | 62.0 (47.24) | 58.8 (46.78)
Statistical Analysis 1: Comparison: Provider-level Push Report Notifications vs No Intervention; Test type: Superiority; p = 0.010, Two-part regression model

ADVERSE EVENTS:
Time Frame: 5 months during which the prescribing for each participant was assessed
Arm/Group | Provider-level Push Report Notifications | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/122
Other Adverse Events (participants affected / at risk) | 0/95 | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT04776928/Prot_000.pdf